CLINICAL TRIAL: NCT06484985
Title: An Open-label, Multicenter, Phase I Safety Study of AXT-1003 in Subjects With Advanced Malignant Tumors
Brief Title: Study of AXT-1003 in Subjects With Advanced Malignant Tumors.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Axter Therapeutics (Beijing) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AXT1003-1102
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Non-Hodgkin Lymphoma; Advanced Solid Tumor
Keywords: AXT-1003; EZH2; Phase I; Advanced malignancies
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AXT-1003 (Experimental): Dose Escalation: Part A:
  Level 1 (Starting Dose) Oral AXT-1003 5 mg BID; Level 2 Oral AXT-1003 10mg BID; Level 3 Oral AXT-1003 15mg BID ; Level 4 Oral AXT-1003 20mg BID; Level 5 Oral AXT-1003 25mg BID; Level 6 Oral AXT-1003 30mg BID; Level 7 Oral AXT-1003 35mg BID; Level 8 Oral AXT-1003 40mg BID;
  Dose Escalation: Part B:
  Oral AXT-1003 2.5mg QD, 10mg BID;
  Dose Expansion: 1 or 2 cohorts at the dose levels selected from dose escalation part
  Interventions: Drug: AXT-1003

INTERVENTIONS:
Drug: AXT-1003 — AXT-1003 capsule is administered orally daily, until disease progression or intolerable toxicity.

SUMMARY:
This is a Phase I study of AXT-1003 to assess the safety, tolerability, and pharmacokinetics in patients with advanced malignancies.

DETAILED DESCRIPTION:
AXT1003-1102 is a multicenter, open-label, Phase I safety study of AXT-1003 in patients with advanced malignancies. It is designed to observe the safety of AXT-1003 in patients with advanced malignancies, determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D), evaluate the pharmacokinetic profile, and explore the preliminary antitumor activity.

ELIGIBILITY:
Inclusion Criteria:

1. For Ia dose escalation part only:

   R/R NHL: Locally histopathological diagnosis of relapsed/refractory non-Hodgkin lymphoma (R/R NHL), who have progressed or been intolerant after the available standard therapies, or have no access to the standard therapies.

   Advanced solid tumors: Locally histopathological diagnosis of locally advanced unresectable and metastatic solid tumors,The above subjects have progressed or been intolerant after the available standard therapies, or have no access to the standard therapies.

   For Ib dose expansion part only: Subjects with relapsed/refractory peripheral T-cell lymphoma (R/R PTCL)
2. Eastern Cooperative Oncology Group (ECOG) performance status scale 0 to 1.
3. Have a life expectancy of at least 3 months.
4. For Ib dose expansion part and not mandatory for Ia dose escalation part: Subjects with R/R NHL must have measurable lesions as defined by Lugano 2014 criteria. Subjects with advanced solid tumors must have measurable or evaluable lesions as defined by RECIST 1.1.
5. Adequate organ and bone marrow functions.
6. The adequate washout period for prior therapy .
7. Subjects must use a highly effective contraception method throughout the study and for 3 months after discontinuation of the study drug.
8. Signed ICF and willing to comply with all the requirements in the protocol.

Exclusion Criteria:

1. Diagnosis of precursor B-cell lymphoblastic leukemia/lymphoma, precursor T-cell lymphoblastic leukemia/lymphoma, precursor NK cell lymphoblastic leukemia/lymphoma. Diagnosis of chronic lymphocytic leukemia (CLL), small lymphocytic lymphoma (SLL).
2. Central nervous system infiltration.
3. Uncontrolled or significant cardiovascular disease.
4. Major surgery within 4 weeks before the first dose of study drug.
5. Known or suspected hypersensitivity to AXT-1003 or any of the excipients.
6. Inability to take oral medication, or malabsorption syndrome or any other uncontrolled gastrointestinal condition (e.g., nausea, diarrhea, or vomiting) that might impair the bioavailability of AXT-1003.
7. History of other malignancies prior to enrollment; except for subjects with basal cell carcinoma of skin, squamous cell carcinoma of skin, cervical carcinoma in situ, or other carcinomas in situ who have undergone possible curative treatment and do not have disease recurrence within 5 years since starting the treatment.
8. Any prior treatment-related clinically significant toxicities that have not resolved to Grade ≤ 1 or prior treatment-related toxicities that are clinically unstable and clinically significant at time of enrollment.
9. Active infection requiring systemic treatment.
10. Infection with hepatitis B virus with positive hepatitis B surface antigen, or hepatitis C virus with detectable anti-hepatitis C circulating viral RNA.
11. Subjects known to be infected with human immunodeficiency virus and active tuberculosis.
12. Females who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Dose-Limiting Toxicity (DLT) (Dose Escalation) | Up to 28 days
  Dose Escalation only: to characterize the dose limiting toxicities (DLTs) of AXT-1003.
Number of Participants with Adverse Events (AEs) | Baseline up to 30 days after the last dose of study
  Laboratory test ,ECG, vital signs, physical examination

SECONDARY OUTCOMES:
Overall response rates (ORR) | Up to 3 years
  ORR is defined as the proportion of subjects with a CR or PR.
Duration of response(DOR) | Up to 3 years
  DOR is defined as the time from the initial objective response to progression of disease (PD) or death after the response, whichever occurs first.
Progression free survival (PFS) | Up to 3 years
  Progression-free survival is defined as the time from the first dose of study treatment to the first PD or death for any reason in the absence of documented PD, whichever occurs first.
Time to response (TTR) | Up to 3 years
  Time to response is defined as the time from first dose of study treatment to the first objective tumor response.
Disease control rate (DCR) | Up to 3 years
  Disease control rate is defined as the proportion of subjects with a CR, PR, or stable disease(SD).
Maximum observed concentration (Cmax) of AXT-1003 | Up to 15 days
  Pharmacokinetics of AXT-1003
Time of maximum observed concentration (tmax) of AXT-1003 | Up to 15 days
  Pharmacokinetics of AXT-1003
Area under the curve from the time of dosing to the time of the last measurable concentration (AUCtau) of AXT-1003 | Up to 15 days
  Pharmacokinetics of AXT-1003
Minimum observed concentration (Cmin) of AXT-1003 | Up to 15 days
  Pharmacokinetics of AXT-1003
Terminal elimination half-life (t1/2) of AXT-1003 | Up to 15 days
  Pharmacokinetics of AXT-1003
Total body clearance (CL/F) of AXT-1003 | Up to 15 days
  Pharmacokinetics of AXT-1003

CONTACTS AND LOCATIONS:
Overall Officials: Qian Gao, Study Director — Axter Therapeutics (Beijing) Co., Ltd
Locations (5):
- China (5):
  - Beijing Cancer Hospital, Beijing
  - Hunan Cancer Hosptial, Changsha
  - Fujian Cancer Hospital, Fuzhou
  - Sun Yat-Sen University Cancer Center, Guangzhou
  - Fudan University Shanghai Cancer Center, Shanghai

IPD SHARING:
Plan to Share IPD: No